CLINICAL TRIAL: NCT04755270
Title: The Effect of Virtual Reality-Supported Hypnofertility on Fertility Preparedness, Stress and Coping With Stress in Women Having In Vitro Fertilization
Brief Title: Virtual Reality-Supported Hypnofertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Çiğdem Erdemoğlu, Research Assistant, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AdıyamanU
Record Dates: First submitted 2021-01-24; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Fertilization in Vitro
Keywords: in vitro fertilization; hypnofertility; stress

STUDY DESIGN:
Intervention Model Description: This research was conducted with the randomized control group pretest-posttest trial model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vr-supported hypnofertility (Experimental): Relaxation, visualization, imagination and affirmation and techniques based on the hypnofertility philosophy were applied to women in the experimental group in four stages
  Interventions: Device: VR Glasses
- Control (No Intervention): Any initiative was not applied to the control group

INTERVENTIONS:
Device: VR Glasses — techniques of hypnofertility and VR glasses
  Other Names: techniques of hypnofertility
  Arms: vr-supported hypnofertility

SUMMARY:
This research was conducted to determine the effect of virtual reality-supported hypnofertility on fertility preparedness, stress and coping with stress in women having in vitro fertilization. At the end of research It has been determined that initiatives based on the hypnofertility philosophy increase the level of preparedness to fertility, decrease the stress level and provide effective coping with stress in women who had IVF treatment.

DETAILED DESCRIPTION:
It is estimated that the infertility affects 8-12% of all couples in reproductive age across the world. Various alternative methods were implemented for years for alleviating the stress which was felt by infertile women. The women in the process of infertility treatment make more efforts to be impregnated, their fertility preparedness is negatively affected and they need more psychosocial support. Upon the review of the relevant literature, it is discerned that there was a limited number of studies in which mind-body programs, namely, hypnofertility methods, were applied to the cases of infertility. In this research, in the first meeting with infertile women who would be assigned to the experimental group, the research objective was explained, and their consent to partake in the research was received in written and verbal format and pretest data were obtained. Later during in vitro fertilization, VR-supported hypnofertility treatment initiative which applied to the experimental group was implemented in four stages, namely, 'Stage 1 (the first folliculometry day)', 'Stage 2 (the second folliculometry day)', 'Stage 3 (oocyte retrieval stage)' and 'Stage 4 (embryo transfer stage)'. And posttest data were obtained at the end of last stage. Each process took 20 minutes on average. Meetings with infertile women who were assigned to the control group were held twice. In the first meeting, pretest data were collected. VR-supported hypnofertility treatment initiative was not applied to the control group, and posttest data were collected from the control group via the second meeting held on the same date as the fourth stage of treatment, namely, the day of embryo transfer. It is considered that the stress levels of women who are in the process of having IVF treatment will fall down and hence the fertility preparedness and the ability to cope with infertility stress will be positively affected by virtue of the effective use of hypnofertility method, which is still a new method in Turkey, by midwives and other health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Having IVF treatment

Exclusion Criteria:

* Having IVF treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Fertility Preparedness Scale for Women Receiving Fertility Treatment | Day 12
  The scale is used for the assessment of the levels of stress experienced by infertile couples. As a Likert-type scale, it has three sub-scales in relation to personal, marital and social domains and contains a total of 14 items. 'Stress in personal domain' sub-scale contains six items, and the minimum and maximum scores to be obtained from it are successively 0 and 20 points. 'Stress in marital domain' sub-scale has four items, and the minimum and maximum scores to be obtained from it are successively 0 and 14 points. 'Stress in social domain' sub-scale is comprised of four items, and the minimum and maximum scores to be obtained from it are successively 0 and 12 points. A high score to be obtained from the sub-scale refers to the increase in the stress level.
The Copenhagen Multi-centre Psychosocial Infertility Fertility Problem Stress | Day 12
  The scale is used for the assessment of the levels of stress experienced by infertile couples. As a Likert-type scale, it has three sub-scales in relation to personal, marital and social domains and contains a total of 14 items. 'Stress in personal domain' sub-scale contains six items, and the minimum and maximum scores to be obtained from it are successively 0 and 20 points. 'Stress in marital domain' sub-scale has four items, and the minimum and maximum scores to be obtained from it are successively 0 and 14 points. 'Stress in social domain' sub-scale is comprised of four items, and the minimum and maximum scores to be obtained from it are successively 0 and 12 points. A high score to be obtained from the sub-scale refers to the increase in the stress level.
The Copenhagen Multi-centre Psychosocial Infertility Coping Strategy Scale | Day 12
  The scale contains 19 items and has four sub-scales. The minimum and maximum scores to be obtained from the sub-scale of 'active-avoidance' coping method which is comprised of four items are successively 4 and 16 points. The sub-scale of 'active-confronting' coping method contains seven items. The minimum and maximum scores to be obtained from this sub-scale are successively 7 and 26 points. The minimum and maximum scores to be obtained from the sub-scale of 'passive-avoidance' coping method which is comprised of three items are successively 3 and 12 points. The sub-scale of 'meaning-based' coping method contains five items. The minimum and maximum scores to be obtained from this sub-scale are successively 5 and 20 points. A higher score to be obtained from the subscale means that the method is used more when coping with with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Aksoy Derya, Phd, Study Director — Inonu University
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers. Because the institution where the research was conducted does not allow this.

REFERENCES:
- [Derived] Erdemoglu C, Aksoy Derya Y. The effect of hypnofertility on fertility preparedness, stress, and coping with stress in women having in vitro fertilization: A randomized controlled trial. J Reprod Infant Psychol. 2024 Jul;42(4):569-580. doi: 10.1080/02646838.2022.2156488. Epub 2022 Dec 13. PMID 36513620